CLINICAL TRIAL: NCT05118061
Title: StatStrip Glucose/Ketone Meter System Ketone Evaluation
Status: Completed | Type: Observational
Sponsor: Nova Biomedical (Industry)
Collaborators: Ocean Wellness Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: NB21-SSK-NA-FDA
Record Dates: First submitted 2021-07-28; First posted 2021-11-11 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Diabetes Mellitus; Ketosis, Diabetic
Keywords: Ketone
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Ketoacidosis; Ketosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Ketone — compare diagnostic tests to reference methods

SUMMARY:
The Nova StatStrip Glucose / Ketone Meter System is a fast, simple, whole blood system that can be used to quantify both glucose and ketones using two distinct test strips. This Protocol will describe an evaluation of the system's Ketone performance only. Ketone testing methods that quantify beta-hydroxybutyrate (β-OHB), the predominant ketone body, are used for diagnosing and monitoring ketoacidosis, a life-threatening complication of hyperglycemia. The performance of the StatStrip Ketone test strip using the Nova StatStrip Glucose / Ketone Hospital Meter System on venous and capillary whole blood will be assessed.

DETAILED DESCRIPTION:
The primary objectives of this study are:

1. To assess the performance of the StatStrip Ketone assay in the hands of CLIA-Waived Point-of-Care users in at least three (3) distinct Point-of-Care clinical settings on venous, and capillary blood and compare the performance characteristics to a traceable laboratory reference method.
2. To assess the Ease of Use of the StatStrip Glucose / Ketone Meter System in the hands of the intended CLIA-Waived Point-of-Care users. CLIA-Waived operators will be provided with all package-insert sheets, a Quick Reference Guide and Instructions for Use (IFU) Manual. No training, coaching, or prompting will be provided to the CLIA-Waived POC Users other than clarifying the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects (≥ 18 years old) with diabetes or suspected ketonemia.
2. Adult subjects (≥ 18 years old) that are healthy.
3. Subjects willing and able to consent to participating in the study.
4. Subjects whose pre-screen ketone value, if performed, is deemed valuable to the study.

Exclusion Criteria:

1. Subjects unable to consent to participating in the study.
2. Subjects possessing a cognitive disorder or other condition, which, in the opinion of the investigator, would put the person at risk or seriously compromise the integrity of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: a minimum of 360 to a maximum of 500 individual subjects will be enrolled to test both capillary and venous whole blood. Subjects included in the study may be healthy, diabetic or suspected of ketonemia. The study will be conducted in at least three (3) separate study sites, with each site targeting 120 patients up to 200 patients.
  Adult subjects (≥ 18 years old) of both genders will be included in this study.
  Potential subjects may be screened prior to testing to assess their baseline ketone levels. The screening may be done by inspecting medical records, fingerstick ketone testing or urine dipstick testing. Each site shall follow their own specified procedures and protocols for the screening test method, if applicable.
Sampling Method: Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Analytical verification of StatStrip glucose/ketone meter system - ketone comparison | 20 days
  StatStrip ketone meter system, a point of care testing instrument is as effective as a reference laboratory method for ketone results in mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Bleicher, MD, Principal Investigator — South Florida Research Organization; Peter Luppa, Principal Investigator — Technical University of Munich
Locations (3):
- South Florida Research Organization, Medley, Florida, United States
- Germany (2):
  - Technical University of Munich - Diabetes Hospital, Munich
  - Technical University of Munich - Emergency Reception, Munich

IPD SHARING:
Plan to Share IPD: No